CLINICAL TRIAL: NCT03375411
Title: INCSTENT First-in-Man Study: Safety and Efficacy of INC-1 Bare Metal Stent in the Novo Coronary Lesions.
Brief Title: First-in-Man Study: Safety and Efficacy of INC-1 Bare Metal Stent in the Novo Coronary Lesions.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: CHANGE TO ANOTHER PLATFORM IN STUDY.
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: GSE Biomedical (Other); Medstent SA de CV. (Unknown)
Responsible Party: Principal Investigator, Gian Manuel Jiménez Rodríguez, Clinical investigator assistant, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-1036
Record Dates: First submitted 2017-10-30; First posted 2017-12-18 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Stents; Coronary Artery Disease; Angioplasty; Humans; Coronary Angiography; Angioplasty, Balloon, Coronary; Treatment Outcome
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INC1-Bare metal stent (Experimental): Percutaneous coronary implantation of the device (Stent INC-1) following the standard procedure of stent placement
  Interventions: Device: Stent INC1

INTERVENTIONS:
Device: Stent INC1 — Coronary intervention with conventional angioplasty technique but with a novel bare metal stent.

SUMMARY:
This is a First In Man study with the aim to know the safety and effectiveness of a novel bare metal stent (INC-1) in the treatment of de novo coronary lesions in patients with stable coronary angina and unique coronary lessions.

DETAILED DESCRIPTION:
The cost of performing a percutaneous coronary intervention is very variable since a large number of materials and human resources are considered, with the Stent cost being a fundamental factor; in developing countries, the cost this technology represents an important expense for the patient and the health system; which promotes the development of local technology to support the requirement of these devices.

Ischemic heart disease together with cerebral vascular events is the main cause of, adding 15 million deaths per year. Percutaneous revascularization is the gold standard choice in many of the variants of presentation of ischemic heart disease, the implantation of Stents is the most used method.

Nowadays more and more countries start their own research and development of novel devices in order to reduce cost.

Research question: Is the INC1 Bare Metal Stent safe and effective for the treatment of de novo coronary lesions in humans? Hypothesis: The INC1 Bare-metal Stent is safe and effective for the treatment of de novo coronary lesions in humans

The INC1 Bare metal Stent is a 70uCoCr

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* From 18 to 75 years
* Stable ischemic heart disease.
* Live less than 300 km from the Institution
* Single coronary artery disease with a single coronary lesion
* Stenosis of 50 to 90% of the lumen of the vessel to be treated.
* Lesions less than 20 mm long
* Reference lumen of the vessel to be treated greater than 2.5mm and less than 4.5mm

Exclusion Criteria:

* Left main disease.
* Lesions greater than 90% of the lumen.
* Non-dilatable lesion with conventional balloons.
* Contraindication for dual antiplatelet therapy.
* Creatinine clearance less than 45ml / min.
* Calcification from moderate to severe.
* Multivessel coronary artery disease.
* Chronic total occlusion.
* Cardiogenic shock or hemodynamic instability.
* Left ventricular ejection fraction less than 30%.
* Valvular disease of moderate to severe.
* Coronary disease in bifurcation.
* Probable or definite presence of thrombus in the lesion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-30 (Estimated); Primary Completion 2018-11-15 (Estimated); Study Completion 2019-01-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of late lumen loss [Safety and Tolerability]) | 9 months
  The primary endpoint of the study is angiographic in-stent late lumen loss (LLL), defined as the difference between the post-procedural minimal lumen diameter (MLD) in the stented segment and the MLD in the same segment at follow-up measured by the angiography laboratory.

SECONDARY OUTCOMES:
Need of Revascularization | 9 months
  The Need of Revascularization of the treated vessel with a new angioplasty
MACE | 9 months
  To evaluate the presence of major adverse cardiovascular events such (MACE) as cardiac death, myocardial infarction, new angina event or revascularization through surgery.
Hyperplasia | 9 months
  To evaluate the degree of neointimal hyperplasia or at 9 months by intracoronary ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Manuel Jiménez Rodríguez, Principal Investigator — Interventional Cardiology
Locations (1):
- Instituto Nacional de Cardiología, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No